Version No.: 2.0

Version Date: 5 January 2023

## INFORMED CONSENT FORM

Title of Study: Phase II Randomized Controlled Trial Of Dendritic Cell + Cytokine-Induced Killer Cell Immunotherapy With S-1 Versus S-1 Alone As Maintenance Therapy For Advanced Pancreatic Ductal Adenocarcinoma Patients (DECIMATE 3.0)

By signing below, I confirm the following:

- I have been given oral and written information for the above study and have read and understood the information given.
- I have sufficient time to consider participation in the study and have had the opportunity to ask questions and all my questions have been answered satisfactorily.
- I understand that my participation is completely voluntary, and I can withdraw anytime from the study without giving a reason and this will in no way affect my future treatment. I am not taking part in any other research study at this time. I understand the risks and benefits, and I freely give my informed consent to participate under the conditions stated. I understand that I must follow the study doctor's (investigator's) instructions related to my participation in the study.
- I understand that study staff, qualified monitors and auditors, the sponsor or its affiliates, and governmental or regulatory authorities, have direct access to my medical record in order to make sure that the study is conducted correctly, and the data are recorded correctly. All personal details will be treated as STRICTLY CONFIDENTIAL.
- I will receive a copy of this subject information/informed consent form signed and dated to bring home.
- I agree/disagree for my family doctor to be informed of my participation in this study.

| Subject: | |
|--------------------------------------------------|-------------|
| Signature: | I/C number: |
| Name: | Date: |
| <b>Investigator conducting informed consent:</b> | 1 |
| Signature: | I/C number: |
| Name: | Date: |

| Version Date: 5 January 2023 | |
|---|---|
| Impartial witness: (Requorally communicated to su | red if subject is illiterate and contents of patient information sheet is<br>bject) |
| Signature: | I/C number: |

Date:

Version No.: 2.0

Name: